CLINICAL TRIAL: NCT02238639
Title: Efficacy and Safety of an Active Strategy for the Diagnosis and Treatment of Acute Pulmonary Embolism (PE) in Patients With Unexplained Exacerbations of Chronic Obstructive Pulmonary Disease (COPD): a Randomized Clinical Trial
Brief Title: Pulmonary Embolism as a Cause of COPD Exacerbations
Acronym: SLICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Spain (Other Government)
Collaborators: American College of Chest Physicians (Other); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, David Jimenez, Senior Consultant, Ministry of Health, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLICE 1
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Embolism; Chronic Obstructive Pulmonary Disease
Keywords: Venous thromboembolism; COPD exacerbations; Anticoagulation; Mortality
MeSH Terms: conditions — Pulmonary Embolism; Pulmonary Disease, Chronic Obstructive; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active search for pulmonary embolism (Experimental): All included patients will undergo D-dimer testing. A negative plasma highly sensitive D-dimer value (defined as a D-dimer level below the manufacturers assay threshold) will rule out pulmonary embolism, and no further examination will be performed. For patients with a positive D-dimer value, a multidetector computed tomographic pulmonary angiography (MDCT) will be performed.
  Interventions: Procedure: Diagnostic and therapeutic strategy: Highly sensitive D-dimer testing and, if positive, multidetector computed tomographic pulmonary angiography (MDCT).
- Standard management (No Intervention): All included patients will undergo standard clinical management of their exacerbations, as deemed appropriate by the attending physician.

INTERVENTIONS:
Procedure: Diagnostic and therapeutic strategy: Highly sensitive D-dimer testing and, if positive, multidetector computed tomographic pulmonary angiography (MDCT). — If MDCT is positive for pulmonary embolism, patients will receive anticoagulant treatment according to updated guidelines.
  If MDCT is negative for pulmonary embolism, patients will receive standard management for their exacerbation.
  Arms: Active search for pulmonary embolism

SUMMARY:
The primary objective is to demonstrate the clinical benefits of an active strategy for the diagnosis and treatment of PE compared to usual care in patients with unexplained exacerbations of COPD who require hospital admission.

The secondary objective is to assess the safety of an active strategy for the diagnosis and treatment of PE compared to usual care in patients with unexplained exacerbations of COPD who require hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of COPD according to SEPAR-ALT criteria: post-bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) < 0.7;
* Hospital admission because COPD exacerbation without initial clinical suspicion of PE in the Emergency Department (according by the Emergency Department physician evaluation).

Exclusion Criteria:

* Contraindication to multidetector computed tomographic angiography (allergy to intravenous contrast medium, or renal failure defined as a creatinine clearance less than 30 mL/min, according to the Cockcroft-Gault formula)
* Informed consent denied
* Pregnancy
* Life expectancy less than 3 months
* Anticoagulant therapy at the time of hospital admission
* Diagnosis of pneumothorax, or pneumonia (fever, and purulent sputum, and new infiltrate in chest X-ray)
* Diagnosis of lower respiratory tract infection (fever [>37.8ºC], increased sputum volume and/or increased sputum purulence).
* Indication of invasive mechanical ventilation at the time of hospital admission;
* Impossibility for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jimenez, MD, PhD, Study Chair — IRYCIS, Alcala de Henares University; Alvar Agusti, MD, PhD, Study Chair — Hospital Clinic; Manuel Monreal, MD, PhD, Study Chair — Germans Trias i Pujol Hospital; Remedios Otero, MD, PhD, Study Chair — Hospital Virgen del Rocio
Locations (19):
- Spain (19):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital La Coruña, A Coruña
  - Hospital Galdakao, Barakaldo
  - Clinica Nostra Senyora del Remei, Barcelona
  - Hospital Capio Sagrat Cor, Barcelona
  - Hospital Cruces, Bilbao
  - Hospital San Pedro, Logroño
  - Hospital Ramon y Cajal, IRYCIS, Alcala de Henares University, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Alcorcon, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital La Paz, Madrid
  - Complejo Hospitalario Pontevedra, Pontevedra
  - Hospital Marques de Valdecilla, Santander
  - Policlinico La Rosaleda, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Peces-Barba G, Barbera JA, Agusti A, Casanova C, Casas A, Izquierdo JL, Jardim J, Lopez Varela V, Monso E, Montemayor T, Viejo JL. [Diagnosis and management of chronic obstructive pulmonary disease: joint guidelines of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) and the Latin American Thoracic Society (ALAT)]. Arch Bronconeumol. 2008 May;44(5):271-81. No abstract available. Spanish. PMID 18448019
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Camargo CA Jr, Roberts J, Clark S. US emergency department visits for COPD exacerbations between 1992 and 1998. Am J Epidemiol 2001; 153: S80.
- [Background] Poulsen SH, Noer I, Moller JE, Knudsen TE, Frandsen JL. Clinical outcome of patients with suspected pulmonary embolism. A follow-up study of 588 consecutive patients. J Intern Med. 2001 Aug;250(2):137-43. doi: 10.1046/j.1365-2796.2001.00866.x. PMID 11489063
- [Background] Tillie-Leblond I, Marquette CH, Perez T, Scherpereel A, Zanetti C, Tonnel AB, Remy-Jardin M. Pulmonary embolism in patients with unexplained exacerbation of chronic obstructive pulmonary disease: prevalence and risk factors. Ann Intern Med. 2006 Mar 21;144(6):390-6. doi: 10.7326/0003-4819-144-6-200603210-00005. PMID 16549851
- [Background] Rizkallah J, Man SFP, Sin DD. Prevalence of pulmonary embolism in acute exacerbations of COPD: a systematic review and metaanalysis. Chest. 2009 Mar;135(3):786-793. doi: 10.1378/chest.08-1516. Epub 2008 Sep 23. PMID 18812453
- [Background] Anderson DR, Kahn SR, Rodger MA, Kovacs MJ, Morris T, Hirsch A, Lang E, Stiell I, Kovacs G, Dreyer J, Dennie C, Cartier Y, Barnes D, Burton E, Pleasance S, Skedgel C, O'Rouke K, Wells PS. Computed tomographic pulmonary angiography vs ventilation-perfusion lung scanning in patients with suspected pulmonary embolism: a randomized controlled trial. JAMA. 2007 Dec 19;298(23):2743-53. doi: 10.1001/jama.298.23.2743. PMID 18165667
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Pozo-Rodriguez F, Lopez-Campos JL, Alvarez-Martinez CJ, Castro-Acosta A, Aguero R, Hueto J, Hernandez-Hernandez J, Barron M, Abraira V, Forte A, Sanchez Nieto JM, Lopez-Gabaldon E, Cosio BG, Agusti A; AUDIPOC Study Group. Clinical audit of COPD patients requiring hospital admissions in Spain: AUDIPOC study. PLoS One. 2012;7(7):e42156. doi: 10.1371/journal.pone.0042156. Epub 2012 Jul 31. PMID 22911875
- [Derived] Najarro M, Briceno W, Rodriguez C, Muriel A, Gonzalez S, Castillo A, Jara I, Rali P, Toma C, Bikdeli B, Jimenez D. Shock score for prediction of clinical outcomes among stable patients with acute symptomatic pulmonary embolism. Thromb Res. 2024 Jan;233:18-24. doi: 10.1016/j.thromres.2023.11.011. Epub 2023 Nov 19. PMID 37988846
- [Derived] Rodriguez C, Muriel A, Carrasco L, Gonzalez S, Briceno W, Duran D, Retegui A, Yusen RD, Bikdeli B, Jimenez D. National Early Warning Score-2 for Identification of Patients with Intermediate-High-Risk Pulmonary Embolism. Semin Thromb Hemost. 2023 Oct;49(7):716-724. doi: 10.1055/s-0043-1769938. Epub 2023 Jun 16. PMID 37327883
- [Derived] Mirambeaux R, Rodriguez C, Muriel A, Gonzalez S, Briceno W, Duran D, Retegui A, Otero R, Bikdeli B, Jimenez D. Comparison of various prognostic scores for identification of patients with intermediate-high risk pulmonary embolism. Thromb Res. 2023 Mar;223:61-68. doi: 10.1016/j.thromres.2023.01.019. Epub 2023 Jan 23. PMID 36708691
- [Derived] Rodriguez C, Jara-Palomares L, Tabernero E, Tenes A, Gonzalez S, Briceno W, Lobo JL, Morillo R, Bikdeli B, Jimenez D. Adjusted D-dimer cutoff levels to rule out pulmonary embolism in patients hospitalized for COPD exacerbation: results from the SLICE trial. Thromb J. 2022 Mar 3;20(1):10. doi: 10.1186/s12959-022-00368-0. PMID 35241119
- [Derived] Jimenez D, Agusti A, Tabernero E, Jara-Palomares L, Hernando A, Ruiz-Artacho P, Perez-Penate G, Rivas-Guerrero A, Rodriguez-Nieto MJ, Ballaz A, Aguero R, Jimenez S, Calle-Rubio M, Lopez-Reyes R, Marcos-Rodriguez P, Barrios D, Rodriguez C, Muriel A, Bertoletti L, Couturaud F, Huisman M, Lobo JL, Yusen RD, Bikdeli B, Monreal M, Otero R; SLICE Trial Group. Effect of a Pulmonary Embolism Diagnostic Strategy on Clinical Outcomes in Patients Hospitalized for COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2021 Oct 5;326(13):1277-1285. doi: 10.1001/jama.2021.14846. PMID 34609451
- [Derived] Jimenez D, Agusti A, Monreal M, Otero R, Huisman MV, Lobo JL, Quezada A, Jara-Palomares L, Hernando A, Tabernero E, Marcos P, Ruiz-Artacho P, Ballaz A, Bertoletti L, Couturaud F, Yusen R; SLICE investigators. The rationale, design, and methods of a randomized, controlled trial to evaluate the efficacy and safety of an active strategy for the diagnosis and treatment of acute pulmonary embolism during exacerbations of chronic obstructive pulmonary disease. Clin Cardiol. 2019 Mar;42(3):346-351. doi: 10.1002/clc.23161. Epub 2019 Feb 25. PMID 30706520

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Search for Pulmonary Embolism: All included patients will undergo D-dimer testing. A negative plasma highly sensitive D-dimer value (defined as a D-dimer level below the manufacturers assay threshold) will rule out pulmonary embolism, and no further examination will be performed. For patients with a positive D-dimer value, a multidetector computed tomographic pulmonary angiography (MDCT) will be performed.
  Diagnostic and therapeutic strategy: Highly sensitive D-dimer testing and, if positive, multidetector computed tomographic pulmonary angiography (MDCT).: If MDCT is positive for pulmonary embolism, patients will receive anticoagulant treatment according to updated guidelines.
  If MDCT is negative for pulmonary embolism, patients will receive standard management for their exacerbation.
Period: Overall Study
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Started | 374 | 372
Completed | 370 | 367
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Search for Pulmonary Embolism | Standard Management | Total
Number analyzed (Participants) | 370 | 367 | 737
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.9) | 70.6 (9.9) | 70.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 109 | 195
  Male | 284 | 258 | 542
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 370 | 367 | 737
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 370 | 367 | 737

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality, Symptomatic Venous Thromboembolism Recurrence, or Need for Readmission.
Description: Clinical composite endpoint of all-cause mortality, or symptomatic venous thromboembolism recurrence, or need for readmission.
Time Frame: 90-day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
Participants | 110 | 107

2. Secondary Outcome: All-cause Mortality
Description: All-cause mortality.
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 23 | 29

3. Secondary Outcome: Symptomatic Recurrent Venous Thromboembolism
Description: Symptomatic venous thromboembolic recurrence confirmed by objective testing.
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 2 | 9

4. Secondary Outcome: Hospitalization
Description: Need for readmission.
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 94 | 84

5. Secondary Outcome: Major Bleeding
Description: Major bleeding (defined according to previously published criteria)
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 3 | 3

6. Secondary Outcome: Clinically Relevant Non Major Bleeding
Description: Clinically relevant non major bleeding (defined according to previously published criteria)
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 1 | 1

7. Secondary Outcome: Serious Adverse Events
Description: Serious adverse events.
Time Frame: 90-day follow-up
Measure: Number; unit: participants
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
Number analyzed (Participants) | 370 | 367
participants | 18 | 18

ADVERSE EVENTS:
Time Frame: 3 months.
Description: Please see protocol.
Arm/Group | Active Search for Pulmonary Embolism | Standard Management
All-Cause Mortality (participants affected / at risk) | 23/370 | 29/367
Serious Adverse Events (participants affected / at risk) | 18/370 | 18/367
Other Adverse Events (participants affected / at risk) | 0/370 | 0/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Search for Pulmonary Embolism (N=370) | Standard Management (N=367)
SAEs (Investigations) | 18 (18) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02238639/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02238639/SAP_001.pdf